CLINICAL TRIAL: NCT00002090
Title: An Open, Multicenter, Randomized, Dose-Ranging Study of Azithromycin in the Treatment of Disseminated Mycobacterium Avium-Intracellulare Complex Infection (MAC) in Patients With Acquired Immune Deficiency Syndrome (AIDS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pfizer (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 058H; 066-148
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1996-04

CONDITIONS: Mycobacterium Avium-Intracellulare Infection; HIV Infections
Keywords: Mycobacterium avium-intracellulare Infection; Acquired Immunodeficiency Syndrome; Azithromycin
MeSH Terms: conditions — Mycobacterium avium-intracellulare Infection; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Azithromycin

INTERVENTIONS:
Drug: Azithromycin

SUMMARY:
To evaluate the efficacy and safety of two doses of azithromycin given chronically for the treatment of Mycobacterium avium bacteremia in AIDS patients.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Medications allowed under a Treatment IND program.

Patients must have:

* HIV infection.
* Disseminated Mycobacterium avium Complex.
* Fever (> 100 degrees F) that cannot be attributed to another active infection, and at least one other constitutional symptom (such as fatigue, malaise, anorexia).
* Life expectancy of at least the duration of the study.
* Consent of parent or guardian if below the legal age of consent.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms and conditions are excluded:

* Known hypersensitivity or significant intolerance to macrolide antibiotics.
* Inability to take oral medications or a current condition likely to interfere with drug absorption (e.g., gastrectomy).

Prior Medication:

Excluded:

* Treatment with an immunostimulant or immunomodulator compound such as alpha-interferon, gamma-interferon, or any interleukin within 7 days prior to study entry.
* Any other antibiotic with known activity against M. avium within 7 days prior to study entry.

Not expected to comply with the requirements of the protocol, in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Beth Israel Hosp, Boston, Massachusetts
  - SUNY / Health Sciences Ctr at Syracuse, Syracuse, New York
  - Bronx Veterans Affairs Med Ctr, The Bronx, New York
  - Ohio State Univ Hosp, Columbus, Ohio
  - United States Air Force Med Ctr, Lackland Air Force Base, Texas
  - Audie L Murphy Veterans Administration Hosp, San Antonio, Texas